CLINICAL TRIAL: NCT01926223
Title: Massachusetts Healthy Families Evaluation-2
Acronym: MHFE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Ann Easterbrooks, Professor, Tufts University
Other Study IDs: TuftsU
Record Dates: First submitted 2013-08-15; First posted 2013-08-20 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Adolescent Parenting
MeSH Terms: interventions — House Calls

ARMS (2):
- Home visiting Group (Experimental)
  Interventions: Other: Home visiting
- Control Group (No Intervention)

INTERVENTIONS:
Other: Home visiting
  Arms: Home visiting Group

SUMMARY:
Massachusetts Healthy Families Evaluation is a randomized controlled trial of a statewide home visiting program for first time parents aged 20 years and under. The evaluation uses a mixed-method design to assess participant outcomes in five program goal areas: 1) prevention child abuse and neglect; 2) optimal child development; 3) educational achievement and economic self-sufficiency; 4) parental well-being; and 5) prevention of repeat teenaged births.

ELIGIBILITY:
Inclusion Criteria:

* age between 16 and 21 years
* first-time parent

Exclusion Criteria:

* cognitive delay
* not fluent in either Spanish or English

Ages: 16 Years to 20 Years | Sex: Female
Age Groups: Child, Adult
Dates: Start 2008-02; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Child abuse and neglect | 24 months post-enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University, Medford, Massachusetts, United States

REFERENCES:
- [Derived] Easterbrooks MA, Bartlett JD, Raskin M, Goldberg J, Contreras MM, Kotake C, Chaudhuri JH, Jacobs FH. Limiting home visiting effects: maternal depression as a moderator of child maltreatment. Pediatrics. 2013 Nov;132 Suppl 2:S126-33. doi: 10.1542/peds.2013-1021K. PMID 24187114